CLINICAL TRIAL: NCT01986283
Title: A Randomized, Double-blind, Triple-dummy, Placebo Controlled, Single-dose, 4-way Crossover Study To Determine The Relative Abuse Potential Of Pf-00345439 (Oxycodone Extended Release Capsules) Compared To Immediate-release Oxycodone And Placebo When Administered Orally Whole And/or Chewed To Non-dependent, Recreational Opioid Users Under Fasted Conditions
Brief Title: Abuse Potential Study of PF-00345439
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B4501016
Record Dates: First submitted 2013-11-01; First posted 2013-11-18 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Opioid Users
Keywords: Abuse potential; PF-00345439; drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Capsules; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Placebo Comparator): Placebo solution +placebo capsule + placebo capsule chewed.
  Interventions: Drug: Capsule
- Treatment B (Experimental): PF-00345439 taken whole + placebo solution + placebo chewed
  Interventions: Drug: PF-00345439
- Treatment C (Experimental): PF-00345439 chewed + placebo solution + placebo taken whole
  Interventions: Drug: PF-00345439
- Treatment D (Active Comparator): Oxycodone HCl immediate-release 40 mg tablets (eg, 2 x 5 mg + 1 x 30 mg) + placebo taken whole + placebo chewed
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: Capsule — Taken once
  Arms: Treatment A
Drug: PF-00345439 — 40 mg capsule swallowed whole, taken once
  Arms: Treatment B
Drug: PF-00345439 — 40 mg capsule chewed, taken once
  Arms: Treatment C
Drug: oxycodone — 40 mg solution, taken once
  Arms: Treatment D

SUMMARY:
This study will determine the relative abuse potential of intact and chewed PF-00345439 (Oxycodone Extended-Release Capsules) compared to crushed oxycodone HCL immediate release (IR) tablets and placebo administered orally to non-dependent, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years who are recreational opioid users and are NOT dependent on opioids.

Exclusion Criteria:

* Evidence or history of clinically significant medical conditions.
* Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine).
* Has participated in, is currently participating in, or is seeking treatment for substance-and/or alcohol-related disorders (excluding nicotine and caffeine).
* Has a positive urine drug screen (UDS) excluding tetrahydrocannabinol (THC).
* Has a positive alcohol breath test.
* Has any history of a condition in which an opioid is contraindicated.
* History of sleep apnea in the past 5 years that has not been resolved or corrected.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results .
* Positive test for Hepatitis B, Hepatitis C, or HIV.
* Allergy or history of hypersensitivity to naloxone HCl, oxycodone HCl, other opioids, and/or lactose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Drug Liking: Peak Effect (Emax) | 12 hours
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS); where 0 mm = Not at all and 100 mm = Extremely.
High: Peak Effect (Emax) | 12 hours
  High assesses the degree that a subject feels a good effect (ie euphoria) at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar scale); where 0 mm = Not at all and 100 mm = Extremely.
Drug Liking: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS); where 0 mm = Not at all and 100 mm = Extremely.
High: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  High assesses the degree that a subject feels a good effect (ie euphoria) at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar scale); where 0 mm = Not at all and 100 mm = Extremely.

SECONDARY OUTCOMES:
Take Drug Again Effect at 24 Hours | 24 hours
  Take drug again visual analogue scale (VAS) is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = Definately not and score of 100 mm = Definately so).
Overall Drug Liking | 24 hours
  Overall Drug Liking visual analogue scale (VAS) is a subjective assessment of the degree to which a participant likes the drug overall. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = Not at all and 100 mm = Extremely).
Any Drug Effects: Area Under Drug Effect Curve (AUE) From 0-1 Hour | 1 hour
  Any drug effects effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Pupillometry: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Chewing Duration | 5 min
  Chewing duration is a measurement of the total time a person is able to chew.
Taste: Subjective Experience from Chewing | 5 min
  Subjective Experience from Chewing is a visual analogue scale (VAS) subjective assessment of the taste of the substance being chewed. Participants are asked to describe the taste of the drug using a VAS with score ranging from 0 mm to 100 mm (score of 0 mm = Extremely unpleasant, 50 mm = neutral, and 100 mm = Extremely pleasant).
Any Drug Effects: Area Under Drug Effect Curve (AUE) From 0-2 Hours | 2 hours
  Any drug effects effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Any Drug Effects: Area Under Drug Effect Curve (AUE) From 0-3 Hours | 3 hours
  Any drug effects effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Any Drug Effects: Area Under Drug Effect Curve (AUE) From 0-12 Hours | 12 hours
  Any drug effects effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Pupillometry: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Pupillometry: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Pupillometry: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
High: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
High: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
High: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Good Drug Effects: Area Under Drug Effect Curve (AUE) From 0-1 Hour | 1 hour
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Good Drug Effects: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Good Drug Effects: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Good Drug Effects: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Bad drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hour
  Bad drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Bad drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Bad drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Feeling Sick: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Feeling sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Feeling Sick: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Feeling sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Feeling Sick: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Feeling sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Feeling Sick: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Feeling sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Nausea: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Nausea: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Nausea: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Nausea: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Sleepy: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Sleepy: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Sleepy: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Sleepy: Area Under Effect Curve (AUE) From 0-12 Hour | 12 hours
  Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Dizzy: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-1).
Dizzy: Area Under Effect Curve (AUE) From 0-2 Hours | 2 hours
  Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-2).
Dizzy: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-3) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-3).
Dizzy: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Bad Effects: Peak Effect (Emax) | 12 hours
  Bad effects visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Nausea: Peak Effect (Emax) | 12 hours
  Nausea visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Feel Sick: Peak Effect (Emax) | 12 hours
  Feel sick visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Sleepy: Peak Effect (Emax) | 12 hours
  Sleepy visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Dizzy: Peak Effect (Emax) | 12 hours
  Dizzy visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Pupillometry: Peak Effect (Emax) | 12 hours
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions.
Good Drug Effects: Peak Effect (Emax) | 12 hours
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-12).
Drug Liking: Area Under Effect Curve (AUE) From 0-1 Hour | 1 hour
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS), where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Drug Liking: Area Under Effect Curve (AUE) From 0-3 Hours | 3 hours
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS), where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Drug Liking: Area Under Effect Curve (AUE) From 0-12 Hours | 12 hours
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS), where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Drug Liking: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm unipolar visual analogue scale (VAS), where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
High: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Any Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Any drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Good Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Good drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Bad Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Bad drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Feel Sick: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Nausea: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Sleepy: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Sleepy visual analogue scale (VAS) assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Dizzy: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Pupillometry: Time to Maximum (Peak) Effect (TEmax) | 12 hours
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. TEmax = Time to maximum observed score.
Any Drug Effects: Peak Effect (Emax) | 12 hours
  Any drug effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'not at all' (score of 0 mm) to 'extremely' (score of 100 mm).
Texture: Subjective Experience from Chewing | 5 mins
  Subjective Experience from Chewing is a visual analogue scale (VAS) subjective assessment of the texture of the substance being chewed. Participants are asked to describe the the texture of the drug using a VAS with score ranging from 0 mm to 100 mm (score of 0 mm = Extremely unpleasant, 50 mm = neutral, and 100 mm = Extremely pleasant).
Maximum Observed Plasma Concentration (Cmax) | 24hr
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 24hr
Area under the curve (AUC) | 24hr
Systemic Clearance (CL) | 24hr
volume of distribution (Vd) | 24hr
Half-Life (t1/2) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501016&StudyName=Abuse%20Potential%20Study%20of%20PF-00345439